

# Facultad de Medicina Instituto de Aparato Locomotor y Rehabilitación

# DOCUMENTO DE INFORMACIÓN PARA EL PARTICIPANTE Y FORMULARIO DE CONSENTIMIENTO INFORMADO

El presente formulario de consentimiento informado va destinado a todo estudiante universitario de Valdivia interesado en participar del estudio "Cambios agudos en los niveles plasmáticos de Adiponectina y FGF21 producto de una sesión de HIIT en estudiantes universitarios inactivos físicamente".

Investigadores: Daniela Alvarado, Antonio González, Mª Belén Reyes y Josefa Videla.

Organizado por: Estudiantes de Kinesiología de la Universidad Austral de Chile (UACH).

Patrocinador: Klgo. Sergio Martinéz Huenchullán

Este documento está formado por dos partes:

- Información
- Formulario de consentimiento informado

#### PARTE I: Información

Somos estudiantes de quinto año de Kinesiología UACH y estamos trabajando en nuestro Proyecto de Tesis, el cual busca estudiar algunos efectos metabólicos que produce el ejercicio en estudiantes que son inactivos físicamente. Precisamente deseamos investigar sobre los cambios en los niveles de dos proteínas que se pueden dar producto de la acción del ejercicio físico.

Le entregaremos información y le invitamos a participar en esta investigación. No tiene que decidir hoy si desea participar o no en la investigación. Antes de tomar una decisión, puede hablar con cualquiera de los integrantes, con quien se sienta cómodo sobre el proyecto. Puede que haya algunas palabras que no entienda. Por favor, me detiene según le informo para darme tiempo a explicarle. Si tiene preguntas más tarde, puede preguntarme a mí, al doctor que investiga o a los miembros del equipo.

# **Propósito**

La inactividad física es cuando las personas no cumplen con las recomendaciones mínimas de realización de actividad física espontánea, las cuales son realizar menos de 150 minutos/semana de actividad física de intensidad moderada o menos de 75 minutos/semana de actividad física vigorosa.

Las personas que son inactivas físicamente se predisponen a desarrollar enfermedades metabólicas y cardiovasculares en el futuro. Es por ello que se recomienda realizar ejercicio físico para prevenirlas.

En relación a esto, el ejercicio promueve la producción de moléculas que favorecen un mejor estado de salud, incluso en personas inactivas físicamente. No obstante, no existe tanta claridad en cómo se generan estos beneficios.

Es por esto que, con la realización de esta investigación, estamos buscando determinar si existe alguna relación entre las personas que son inactivas físicamente y el posible aumento de ciertas proteínas a nivel plasmático (en la sangre) antes del ejercicio y posterior a este.

# Tipo de intervención de investigación

Esta investigación incluirá 1 día para reconocer el espacio e implementos que serán ocupados durante la investigación y su participación, además de otro día donde se realizará la sesión de ejercicio; ambas en un día y horario a convenir entre el equipo de investigación y usted.

Antes de comenzar la sesión de ejercicio, se realizarán mediciones de signos vitales además de la toma de muestra de sangre venosa desde su brazo, procedimiento que será ejecutado por alguien entrenado para hacerlo.

La sesión de ejercicio se realizará en treadmill (trotadora), en donde comenzará con cargas bajas las cuales se irán aumentando progresivamente. Posterior a la realización de la sesión de ejercicio, se realizará nuevamente la toma de signos vitales y muestra de sangre a modo de investigar qué cambios ocurrieron con el ejercicio.

# Selección de participantes

Pueden participar todos los estudiantes universitarios de la ciudad de Valdivia que sean inactivos físicamente, cumplan con los criterios de inclusión y que estén interesados en participar.

La selección de participantes por medio de los criterios de inclusión incluye:

- Tener entre 18 a 29 años de edad.
- Sujetos que sean inactivos físicamente, es decir que no cumplan con 150 minutos de AF de intensidad moderada recomendados por la OMS.
- En el cuestionario de PARQ no debe existir ninguna respuesta positiva.

# Participación voluntaria

Su participación en esta investigación es totalmente voluntaria. Usted puede elegir participar o no hacerlo. Tanto si elige participar o no, continuarán todos los servicios que reciba y nada cambiará. Usted puede cambiar de idea más tarde y dejar de participar aun cuando haya aceptado antes.

# **Procedimientos y protocolos**

Como parte de este estudio, le pediremos realizar una prueba física, contestar cuestionarios y además necesitaremos pequeñas muestras de sangre venosa (5 ml). A continuación, se explican las diferentes pruebas:

1. Realización de HIIT: Acá le pediremos que trote en el treadmill, en velocidades establecidas de intervalos de alta intensidad y de baja intensidad, que se irán intercalando entre sí. La prueba finalizará cuando usted finalice con el ciclo establecido de HIIT o bien cuando sea incapaz de seguir. Constantemente se le medirán los signos vitales (pulso, presión arterial, percepción de esfuerzo) para asegurarnos de que está realizando la prueba de manera segura.



- **2. Medidas antropométricas:** Su peso, talla (estatura), junto con su circunferencia (perímetro) de cintura y cadera serán medidas para caracterizar la forma de su cuerpo.
- 3. Composición corporal: Aquí le pediremos que se ubique de pie y tomé un instrumento llamado bioimpedanciómetro, el cual puede medir la cantidad de músculo y grasa que tiene en su cuerpo, de manera indirecta. Acá no sentirá absolutamente nada mientras el instrumento está funcionando. La medición dura 2 a 3 minutos.
- i da
- 4. Actividad física espontánea: Para medir el nivel de actividad física que usted realiza, se le aplicará un cuestionario que relaciona la actividad realizada durante más de 10 minutos en actividades como caminata, actividades moderadas y vigorosas. Además, involucra 4 ámbitos de la actividad física como el trabajo, transporte, actividades del hogar y el tiempo libre. En cada uno se incluye el número de días por semana, tiempo por semana y el tiempo diario dedicado a cada actividad.
- 5. Toma de muestra de sangre venosa: Tanto antes como después de la realización de la sesión de ejercicio, se tomará una muestra de sangre venosa desde su brazo. Con esto se tomarán exámenes de laboratorio para poder identificar los efectos del ejercicio en su persona. Aquí se tomarán dos tubos de sangre, uno con anticoagulante (para obtener plasma) y otro sin anticoagulante (para obtener suero). La cantidad



- de sangre a obtener será de un máximo de 10 ml, o 2/3 de una cucharada sopera. Estas muestras de sangre sólo serán utilizadas para este estudio. Luego de esto serán eliminadas.
- **6.** Medición de glicemia y de lactato sanguíneo: Se valorarán a través de instrumentos portátiles que requieren sólo una gota de sangre desde uno de sus dedos a través de una lanceta estéril.



# Descripción del proceso

Durante el estudio, usted tendrá que asistir 2 veces al Edificio de Ciencias del Movimiento Humano y la Ocupación (ECMHO), ubicado en la calle Rudloff 1650.

La primera visita tiene como propósito, que usted se familiarice con el Laboratorio de Fisiología del Ejercicio y los implementos que serán ocupados durante el transcurso de la intervención, además de esto se le aplicarán una serie de cuestionarios que tienen por finalidad determinar si cumple con los criterios de inclusión establecidos en nuestra investigación, los cuales ya fueron mencionados anteriormente y, por último, se le realizará la medición de composición corporal.

Si cumple con los criterios de inclusión se le pedirá que asista por segunda vez al Laboratorio de Fisiología del Ejercicio, donde, en esta ocasión se le hará la toma de

muestras sanguíneas tanto pre como post sesión de HIIT, toma de signos vitales pre y post y para finalizar se comenzará con la sesión de entrenamiento HIIT qué cuenta, como ya se mencionó, con la toma de signos vitales al finalizar la sesión.

#### Duración

La investigación tendrá una duración total de 1 día. Para ello, será necesario que venga al Edificio de Ciencias del Movimiento Humano y de la Ocupación, en el Laboratorio de Fisiología del Ejercicio. Inicialmente se le aplicaran dos cuestionarios de salud, para confirmar o no su participación. Si estos cuestionarios lo permiten, se continuará con los procedimientos y protocolos ya descritos. Tendrá una duración aproximada de una hora y media.

#### **Efectos secundarios**

Estos procedimientos puede que tengan algún efecto no deseado. Puede que le haga sentirse cansado y puede causar malestar físico o psíquico. Es posible que pueda también causar problemas que no conocemos. Sin embargo, le haremos un seguimiento y mantendremos un registro de cualquier efecto no deseado o cualquier problema.

Si fuera necesario, solicitaremos evaluación médica en caso de encontrarnos con problemas o efectos no deseados. Si esto es necesario lo discutiremos con usted y siempre se le consultará antes de continuar con el próximo paso.

# Riesgo

Al participar en esta investigación es posible que usted se exponga a un riesgo mayor que si no lo hiciera. Existe, por ejemplo, el riesgo de que tenga dolores musculares y/o articulares, asociados a las pruebas o a la sesión de ejercicio físico.

Sin embargo, es esperable y normal que estas molestias comiencen a bajar despues de 48 horas de haber realizado los esfuerzos físicos. Si esto no ocurre, solicitaremos asistencia médica para solucionar sus síntomas de la mejor forma posible.

Además, es posible que aparezcan hematomas en la zona de extracción de las muestras de sangre. Minimizamos esta posibilidad, al contar con profesionales que realicen este procedimiento. Sin embargo, si hubiera complicaciones con este procedimiento, solicitaremos la asistencia médica correspondiente.

# **Molestias**

Al participar en esta investigación, es posible que experimente molestias como el que le tomemos varias veces la presión sanguínea o pincharle las venas. Además de las molestias musculares y articulares asociadas al esfuerzo físico por las pruebas y ejercicio a realizar.

### **Beneficios**

El presente estudio entregará de forma gratuita los resultados de los exámenes de laboratorio que se le tomarán, además de los resultados de la bioimpedancia para composición corporal.

### Incentivos

En este estudio no se contemplan incentivos monetarios para los participantes.

# Confidencialidad

La información que se irá recopilando de usted, que serían sus datos personales, respuestas de cuestionarios pre-participativos, resultados de exámenes de sangre, resultados de composición corporal y de la prueba física, serán totalmente confidenciales.

#### Resultados

Los resultados de su participación se compartirán con usted, antes de que estos datos sean difundidos públicamente al dar a conocer el estudio. No obstante, ninguno de los resultados se compartirán con su identidad o datos personales.

# Derecho a negarse o retirarse

Así como la participación es voluntaria, se recalca que no es obligación participar, incluso si ha iniciado el proceso, puede retirarse en cualquier momento, estando en todo su derecho.

# A quién contactar

Ante cualquier consulta posterior, puede comunicarse con alguno de los investigadores:

**Daniela Alvarado Carrasco** 

Celular: +56933133826

Email: daniela.alvarado02@alumnos.uach.cl

Antonio González Maraboli Celular: +56985431648

Email: antonio.gonzalez@alumnos.uach.cl

Mª Belén Reyes Montalva Celular: +56966128581

Email: maria.reyes02@alumnos.uach.cl

Josefa Videla Aguilar Celular: +56997909072

Email: josefa.videla@alumnos.uach.cl

Dirección: Rudloff 1650, Valdivia.

Este proyecto ha sido revisado y aprobado por el Comité Ético Científico del Servicio de Salud Valdivia. Este Comité está acreditado y tiene como función resguardar los derechos de las personas como sujetos de investigación. Si usted desea averiguar más sobre esté comité, contacte al teléfono: 63-2281784 o en Edificio Prales, Vicente Pérez Rosales 560, oficina 307, 3° piso, Valdivia, Chile.

# PARTE II: Formulación de Consentimiento Informado

- He sido invitado a participar en la investigación sobre los efectos de una sesión de ejercicio sobre marcadores sanguíneos y clínicos en personas inactivas físicamente.
- Entiendo que deberé realizar una sesión de ejercicio físico durante 1 día.
- He sido informado de que los riesgos son mínimos y pueden incluir solo dolor muscular y articular, además de posibles hematomas en las zonas donde se realicen tomas de muestras de sangre.
- Sé que puede que no haya beneficios para mi persona y que no se me compensará más allá de los gastos asociados a los exámenes de laboratorio.

- Se me ha proporcionado el nombre de los investigadores, que pueden ser fácilmente contactados usando el nombre, número de celular, correo electrónico y dirección.
- He leído la información proporcionada o me ha sido leída.
- He tenido la oportunidad de preguntar sobre ella y se me ha contestado satisfactoriamente las preguntas que he realizado.

| Consiento No consiento |
|---|
| voluntariamente participar en esta investigación como participante y entiendo que tengo derecho de retirarme en cualquier momento sin que me afecte en ninguna manera mi cuidado médico. |
| Nombre del participante: |
| Firma del participante: |
| Fecha: (día/mes/año) |
| He leído con exactitud o he sido testigo de la lectura exacta del documento de consentimiento informado para el potencial participante y el individuo ha tenido la oportunidad de hacer preguntas. Confirmo que el individuo ha dado consentimiento libremente. |
| Nombre del investigador: <u>Daniela Carolina Alvarado Carrasco</u> |
| Firma: |
| Fecha: (día/mes/año) |
| Nombre del investigador: Antonio Jonathan Josue González Maraboli |
| Firma: |
| Fecha: (día/mes/año) |
| Nombre del investigador: <u>María Belén Reyes Montalva</u> |
| Firma: |
| Fecha: (día/mes/año) |
| Nombre del investigador: <u>Josefa Andrea Videla Aguilar</u> |
| Firma: |
| Fecha: (día/mes/año) |
| Nombre del Director de Establecimiento, |

Delegado o Ministro de Fe: \_\_\_\_\_

| Filma: | |
|---|---|
| Fecha: | Día/mes/año |
| Ha sido proporcionada al partic | sipante una copia de este documento de Consentimiento |
| Informado (iniciales del inv | restigador/asistente). |